CLINICAL TRIAL: NCT04868721
Title: Evaluation of Two Approaches of Micro-osteoperforations During Orthodontic:A Prospective Clinical Study
Brief Title: Evaluation of Two Approaches of Micro-osteoperforations (MOPs) During Orthodontic Canine Retraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Bassem Atef Hassan Ahmed, Dentist, Ministry of Health-Egypt, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 535/1147
Record Dates: First submitted 2021-04-25; First posted 2021-05-03 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Bimaxillary Protrusion; Angle Class II, Division 1; Dental Malocclusions
Keywords: Micro-osteoperforation; Accelerated orthodontics; Tooth movement; Canine retraction
MeSH Terms: conditions — Malocclusion, Angle Class II | interventions — morpholinopropane sulfonic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control side (No Intervention): Conventional side Canine retraction was commenced without micro-osteoperforations.
- single Micro-osteoperforations side (Experimental): Three flapless micro-osteoperforations (MOPs) was performed for one time only distal to the maxillary canine before starting retraction.
  Interventions: Procedure: micro-osteoperforations
- Multiple Micro-osteoperforations side (Experimental): Three flapless micro-osteoperforations (MOPs) was performed on repeated basis distal to the maxillary canine evey 28 days before canine retraction.
  Interventions: Procedure: micro-osteoperforations

INTERVENTIONS:
Procedure: micro-osteoperforations — three flapless micro-osteoperforations was performed distal to the maxillary canine before starting retraction.
  Other Names: MOPs
  Arms: Multiple Micro-osteoperforations side; single Micro-osteoperforations side

SUMMARY:
The aim of this clinical prospective study will be directed to evaluate two approaches of micro-osteoperforations (MOPs) during orthodontic canine retraction.

DETAILED DESCRIPTION:
The aim of the present clinical study was directed to evaluate the effectiveness of two approaches of micro-osteoperforations (MOPs) during orthodontic canine retraction.

This study was conducted on a total sample of 36 canines of 18 patients, 15-22 years old who required therapeutic extraction of maxillary 1st premolars and canine retraction. They were selected randomly from the Outpatient Clinic, Department of Orthodontics, Faculty of Dental Medicine (Boys), Al-Azhar University, Cairo, Egypt.

they were randamly dived into two groups:as follows: Group I: include 9 patients , MOPs were performed for one time only on one side before retraction.

Group II: include 9 patients , MOPs were performed on repeated basis on one side.

Both maxillary canines, in each patient, were randomly assigned to either an experimental side or the control side in a simple split-mouth design. In the experimental side, micro-osteoperforations was performed distal to the maxillary canine at equal distance between maxillary canine and 2nd premolar before starting retraction, while the canines in the contralateral control side were retracted without micro-osteoperforations.

Extraction was done at the start of the treatment, and before fitting of the orthodontic appliance. Then upper dental arches were leveled and aligned using conventional sequences of wires.

Three flapless micro-osteoperforations was performed by using orthodontic miniscrews distal to the maxillary canines in the experimental side before starting retraction. Each perforation was 1.6 mm in diameter and 3-4 mm depth into the bone. Canines were completely retracted on 0.016 × 0.022 ̋ stainless steel wires by using closed coil spring delivered 150 gm force.

Patients were followed up every 28 days for 4 months of canine retraction. Routine orthodontic records were obtained for each patient before treatment.

Additionally, a full skull CBCT images were taken before treatment and immediately after canine retraction.

The rate of canine retraction was assessed clinically; in addition, cone beam CT (CBCT) scans were used to assess the amount of canine retraction root length changes. Also anchorage loss of first permanent molars were assessed.

The treatment results were compared clinically and radiographically (CBCT).

ELIGIBILITY:
Inclusion Criteria:All patients should satisfy the following criteria:-

1. Age range from 15-22 years.
2. Malocclusion cases that require maxillary first premolars extractions followed by symmetrical canine retraction.
3. All permanent teeth present, 3rd molars are excluded.
4. Good oral and general health.
5. No systemic disease/medication that could interfere with OTM.
6. No previous orthodontic treatment.

Exclusion Criteria:

1. Patient diagnosed to have an indication for non-extraction approach.
2. Poor oral hygiene or periodontally compromised patient.
3. Patient with craniofacial anomalies or previous history of trauma, bruxism or parafunctions.
4. Previous orthodontic treatment.

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Rate of canine retraction | change from start of canine retraction until 4 months .
  clinically, patients were evaluated immediately before canine retraction and every 28days until for months.
  It was based on measuring the distance between the contact points on the distal surface of the canines and the contact points on mesial surface of the second premolars.

CONTACTS AND LOCATIONS:
Locations (1):
- Al azhar university, Cairo, Egypt